CLINICAL TRIAL: NCT00768820
Title: The Psychiatric and Cognitive Phenotypes in Velocardiofacial Syndrome (VCFS), Williams Syndrome (WS)and Fragile X Syndrome Characterization, Treatment and Examining the Connection to Developmental and Molecular Factors
Brief Title: The Psychiatric and Cognitive Phenotypes in Velocardiofacial Syndrome
Acronym: VCFS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Chaim Sheba Medical Center (Other)
Responsible Party: Principal Investigator, Prof. Doron Gothelf, Principal Investigator, The Chaim Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SCMCI082455CTIL
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Velocardiofacial Syndrome; Williams Syndrome; Fragile X Syndrome
Keywords: Velocardiofacial syndrome; Williams syndrome; fragile X syndrome; cognitive phenotype; psychiatric phenotype
MeSH Terms: conditions — DiGeorge Syndrome; Williams Syndrome; Fragile X Syndrome | interventions — Methylphenidate; Fluoxetine; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: methylphenidate, fluoxetin, risperidone

INTERVENTIONS:
Drug: methylphenidate, fluoxetin, risperidone — first cognitive evaluation without methylphenidate,second cognitive evaluation with methylphenidate

SUMMARY:
The purpose of this study is to investigate the Psychiatric and Cognitive Phenotypes in Velocardiofacial Syndrome (VCFS), Williams Syndrome (WS)and Fragile X Syndrome Characterization, Treatment and Examining the Connection to Developmental and Molecular Factors

ELIGIBILITY:
Inclusion Criteria:

* chromosomal deletion proven by FISH examination

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2001-05; Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Measure that are used: psychological measures, molecular tests, responsiveness to medical treatments | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Schneider Children's Mediac Center of Israel, Petah Tikva, Israel